CLINICAL TRIAL: NCT01783899
Title: Clinical Evaluation of Hemospray in Hemostasis of Active Variceal Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Collaborators: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Mostafa Ibrahim, Gastroenterologist, Theodor Bilharz Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hemospray Varices
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Variceal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hemospray Group (Experimental): Hemospray device consists of a syringe containing the Hemospray powder (21 g per syringe), a delivery catheter that will be inserted into the working channel of the endoscope, and an introducer handle with a built-in carbon dioxide canister to propel the Hemospray powder out of the catheter.
  In addition to Hemospray device any other required endoscopic accessories can be used during the procedure.
  Interventions: Device: Hemospray

INTERVENTIONS:
Device: Hemospray — Patients will be resuscitated as needed to achieve hemodynamic stability in preparation for endoscopy within 24 hours of hospital admission.
  once the bleeding point will be identified at endoscopy, the delivery catheter will be inserted through the endoscope and positioned toward the lesion, leaving 1-2 cm between the bleeding site and the catheter tip.
  Hemospray will be then delivered in short spray bursts (for 1-2 seconds) until hemostasis was confirmed.
  Once bleeding was controlled , the bleeding site will be observed for 5 minutes under endoscopy.
  Oral food and fluid will be with held from the patient for 24 hours. Intravenous octreotide and esomeprazole will given for up to 24 hours. Patients will be closely monitored for signs of recurrent bleeding for 24 hours post procedure.
  Recurrent bleeding will be diagnosed any patient experiencing recurrent bleeding will treated according to the institutional standard of care

SUMMARY:
The objective of this study is to assess the effectiveness of Hemospray in achieving initial hemostasis and decreased rate of re-bleeding in patients of acute variceal bleeding.

ELIGIBILITY:
Inclusion criteria :

* 18 Years and older
* Bleeding Esophageal and / or Gastric varices

Exclusion Criteria:

* Patient is: < 18 years of age
* Unable to consent
* Contraindicated to undergo endoscopy,
* Already hospitalized for another illness
* Pregnant or lactating
* Patients with altered post-surgical anatomy of the stomach
* Previously placed intrahepatic portosystemic shunt
* Patient treated by other endoscopic or surgical modalities within 7 days prior to the intended application of Hemospray

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Safety | 24 hours
  Safety will be characterized by the incidence of all Adverse Device Effects (ADEs), non-serious and serious, possibly related to or related to the procedure and/or device that are experienced by study participants.

SECONDARY OUTCOMES:
Effectiveness | 24 hours
  Information on efficacy will be obtained by measurements the proportion of patients with acute (procedural) hemostasis, and the rate of recurrent bleeding within 72 hours of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Ibrahim, MD, Principal Investigator — Université Libre de Bruxelles
Locations (2):
- Erasme Hospital , ULB, Brussels, Belgium
- Theodor Bilharz Research Institute, Giza, Egypt

REFERENCES:
- [Derived] Ibrahim M, El-Mikkawy A, Mostafa I, Deviere J. Endoscopic treatment of acute variceal hemorrhage by using hemostatic powder TC-325: a prospective pilot study. Gastrointest Endosc. 2013 Nov;78(5):769-73. doi: 10.1016/j.gie.2013.07.037. PMID 24120338